CLINICAL TRIAL: NCT01220921
Title: Neurosurgery Patient Outcomes in Treating Spinal Disorders
Acronym: Neuropoint SD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Greenwich Hospital (Other)
Collaborators: American Association of Neurological Surgeons (Other)
Responsible Party: Zoher Ghogawala MD FACS, Wallace Clinical Trials Center - Greenwich Hospital - Yale New Haven Health
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Neuropoint SD
Record Dates: First submitted 2010-10-13; First posted 2010-10-14 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2015-12

CONDITIONS: Symptomatic Lumbar Disc Herniation; Symptomatic Grade I Lumbar Spondylolisthesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lumbar Microdiscectomy (Experimental): Patients aged 18-80 with symptomatic lumbar disc herniation resulting in single nerve root compression recalcitrant to non-invasive therapies for at least 6 weeks
  Interventions: Procedure: Lumbar Discectomy
- Single-Level Lumbar Fusion (Experimental): Patients aged 18-80 with symptomatic grade I degenerative or isthmic spondylolisthesis with mechanical back pain with or without radiculopathy recalcitrant to non-invasive therapies for at least 3 months
  Interventions: Procedure: Single-level lumbar fusion

INTERVENTIONS:
Procedure: Lumbar Discectomy — Microsurgical removal of disc that is compressing a nerve root
  Arms: Lumbar Microdiscectomy
Procedure: Single-level lumbar fusion — pedicle screws with arthrodesis as directed by surgeon. Fusion can be posterolateral, interbody, or both.
  Arms: Single-Level Lumbar Fusion

SUMMARY:
The creation of a multi-center cooperative research group encompassing academic and community-based spinal practices . . .

ELIGIBILITY:
Inclusion Criteria:

* Grade I degenerative or isthmic spondylolisthesis recalcitrant to non-invasive therapies for at least 3 months or Lumbar degenerative disc herniation with radiculopathy refractory to non-invasive therapies for at least 6 weeks

Exclusion Criteria:

* History of previous lumbar spine surgery
* Significant motor weakness (3/5) (i.e. foot drop)
* Cancer, infection, or fracture
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2010-09; Primary Completion 2011-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
SF-36 version 1 | 1-Year
  Health-realted quality of life outcome measure
Site and Physician Compliance | 1 Year
  Goal = 80% compliance in enrolling 20 patients over 1 year with completed outcomes instruments

SECONDARY OUTCOMES:
Oswestry Disability Index (ODI) | 1 Year
  Validated lumbar spine disease-specific outcomes instrument
Visual Analog Pain Score | 1 Year
  Patient-reported pain intensity scored 1-10
Return to Work | 1 Year
  Return to work assessments will be performed at 1,3,6, and 12 months post-operatively
30 day complications | 30 days
  death, myocardial infarction (MI), pulmonary embolism (PE), readmission, wound infection, new neurological deficit, re-operation
Delayed Surgical Complications | 1 year
  re-operation, fusion complication, problems with hardware, deformity

CONTACTS AND LOCATIONS:
Overall Officials: Zoher Ghogawala, MD FACS, Study Director — Yale University
Locations (13):
- United States (12):
  - University of California - San Francisco, San Francisco, California
  - Greenwich Hospital, Greenwich, Connecticut
  - Yale New Haven Hospital, New Haven, Connecticut
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Lahey Clinic, Burlington, Massachusetts
  - University of Medicine and Dentistry - New Jersey, Newark, New Jersey
  - Columbia University - Neurological Institute, New York, New York
  - Carolina Spine, Charlotte, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Virginia, Charlottesville, Virginia
  - University of Wisconsin, Madison, Wisconsin
- University of Calgary - Alberta Health Sevices, Calgary, Alberta, Canada